CLINICAL TRIAL: NCT05717218
Title: Ultra-protective Ventilation Monitored by Electrical Impedance Tomography in Patients With Severe Acute Respiratory Distress Syndrome on Veno-venous ECMO
Acronym: EIT-ECMO
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: APHP230064
Record Dates: First submitted 2023-01-19; First posted 2023-02-08 (Actual); Last update posted 2025-05-15 (Actual); Status verified 2025-05

CONDITIONS: Severe ARDS
Keywords: ECMO; ARDS; ultra-protective mechanical ventilation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Interventional (Experimental): All patients included
  Interventions: Device: Ultra-protective mechanical ventilation monitored by electrical impedance tomography

INTERVENTIONS:
Device: Ultra-protective mechanical ventilation monitored by electrical impedance tomography — A silicone EIT belt will be placed around the patient's thorax (sixth intercostal parasternal space). EIT data will be generated by application of a small alternating electrical current (5 mA at 50 kHz). Introduction of "ultraprotective" mechanical ventilation will be monitored.

SUMMARY:
For ECMO supported patients with severe ARDS (acute respiratory distress syndrome), usual care include use of "ultraprotective" mechanical ventilation with tidal volume and pressure reductions that might ultimately enhance lung protection of patients with ARDS. Although very low tidal might also cause pulmonary derecruitment. The aim of this study is to monitor effects of very low tidal volume on regression of overdistension and derecruitment using electrical impedance tomography.

Secondary aim is to describe the evolution of the optimal PEEP (Positive End Expiratory Pressure) during the decrease of the tidal volume

DETAILED DESCRIPTION:
Patients requiring venovenous ECMO support for severe ARDS will be monitored with electrical impedance tomography during introduction of "ultraprotective" mechanical ventilation.

Monitoring will start with pre-ECMO ventilator setting, then the tidal volume will be lowered step by step. Other parameters of the ventilator will be kept constant. Then, cumulated collapse and overdistention percentages will be estimated for each tidal volume. Optimal tidal volume will be defined by the lowest sum of alveolar overdistension and collapse.

Also, at the end of each step, PEEP titration will be performed to identify the optimal PEEP setting that combines the best alveolar recruitment with minimal overdistention. The aim is to determine whether the derecruitment induced by the decrease in tidal volume can be reduced by the application of PEP. Then, comparison of the different tidal volumes with application of ideal PEEP will be performed: measurement of the percentage of collapsed and overdistended areas by impedancemetry method between the different levels of tidal volume with application of ideal PEEP.

ELIGIBILITY:
Inclusion Criteria:

* aged ≥ 18 years
* patient with ARDS on venovenous (VV)-ECMO
* Written informed consent
* patient affiliated to a social security scheme

Exclusion Criteria:

* Pregnancy
* Adult patient subject to a legal protection measure (tutor, curator, etc.)
* Patients with a pacemaker, automatic implantable cardioverter defibrillator,
* contraindications to thoracic belt placement (e.g., thoracic or spinal cord trauma, recent thoracic surgery)
* undrained pneumothorax, bronchopleural fistula
* hemodynamic instability (i.e., use of intravenous fluids of more than 10 mL/kg or vasopressors 2 mg/h of norepinephrine or 0.5 mg/h of epinephrine)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2023-03-11 (Actual); Primary Completion 2027-03-11 (Estimated); Study Completion 2027-05-11 (Estimated)

PRIMARY OUTCOMES:
cumulated collapse and overdistention percentages for each tidal volume by impedancemetry method | One day
  Estimating the "best" lung-compartment compliance, reflected by the number of functional lung units in that region, and current compliance for each pixel, the collapse and overdistention percentages per pixel will be compared for each tidal volume, with constant (pre-ECMO) PEEP.

SECONDARY OUTCOMES:
Optimal PEEP by impedancemetry method at each tidal volume | One day
  PEEP titration will be performed to identify the optimal PEEP setting that combines the best alveolar recruitment with minimal overdistention at each tidal volume
cumulated collapsed and overdistended for each tidal volume by impedancemetry method with application of optimal PEEP | One day
  Estimating the "best" lung-compartment compliance, reflected by the number of functional lung units in that region, and current compliance for each pixel, the collapse and overdistention percentages per pixel will be compared for each tidal volume, with optimal PEEP

CONTACTS AND LOCATIONS:
Locations (1):
- Service de médecine intensive - réanimation Hopital Pitié Salpêtrière, Paris, France

IPD SHARING:
Plan to Share IPD: No